CLINICAL TRIAL: NCT04211766
Title: Diet and the Colonic Exfoliome: A Novel, Non-Invasive Approach to Testing Interventions in Humans
Brief Title: Fiber and Fish Oil Supplements for the Prevention of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Texas A&M University (Other)
Responsible Party: Principal Investigator, Johanna Lampe, Professor, Fred Hutchinson Cancer Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: RG1006100; NCI-2019-07435 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1006100 (Other: Fred Hutch/University of Washington Cancer Consortium); R21CA245456 (NIH); 10327 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2019-11-20; First posted 2019-12-26 (Actual); Results first posted 2023-10-17 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Healthy Subject
Keywords: Colon; Rectum
MeSH Terms: interventions — Dietary Fiber; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cross-over Randomization 1: Fiber plus Fish Oil followed by Comparator (Experimental): Participants first received a fiber supplement and a fish oil supplement PO daily for 30 days (Period 1). Participants entered a washout period for at least 60 days. For period 2 they received similarly packaged comparator (maltodextrin and corn oil)
  Interventions: Dietary Supplement: Dietary Fiber; Dietary Supplement: Fish Oil; Other: Comparator
- Cross-over Randomization 2: Comparator followed by Fiber plus Fish Oil (Experimental): Participants first received the comparator (maltodextrin and corn oil) supplement PO daily for 30 days (Period 1). Participants enter a washout period for at least 60 days. For period 2 they received the fiber supplement and a fish oil supplement
  Interventions: Dietary Supplement: Dietary Fiber; Dietary Supplement: Fish Oil; Other: Comparator

INTERVENTIONS:
Dietary Supplement: Dietary Fiber — Given fiber supplement
  Other Names: Fiber
Dietary Supplement: Fish Oil — Given fish oil supplement
  Other Names: Oil, Fish; Seafood Oil
Other: Comparator — Given fiber supplement placebo
  Other Names: placebo therapy; PLCB; sham therapy
Other: Comparator — Given fish oil supplement placebo (corn oil)
  Other Names: placebo therapy; PLCB; sham therapy

SUMMARY:
This trial studies how fiber and fish oil supplements affect the metabolism and activities of colon cells in healthy individuals. Diet is an important risk factor for colorectal cancer, and several dietary components important in colorectal cancer prevention are modified by gut microbial metabolism. Giving fiber and fish oil supplements may inhibit the growth of gut cells and ultimately reduce risk of colorectal cancer.

DETAILED DESCRIPTION:
Participants are randomized to receive two dietary interventions in assigned random order. They either receive the dietary fiber supplement and fish oil supplement orally (PO) daily or they receive a fiber control and corn oil supplement daily for 30 days during the first intervention period. Then they enter a washout period for 60 days when they do not receive any treatment. After that they complete the second intervention period during which they receive the other intervention.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Normal-overweight (body mass index [BMI] of 18-30 kg/m^2)
* Women will be postmenopausal, with no menstrual period in 12 months
* Non-smoking
* Consume fiber intakes of less than < 20 g/d
* White blood cell count 3,000-11,000/mm^3
* Platelet count 100,000-400,000 mm^3
* Hematocrit 33-50% (women); 36-50% (men)
* Bilirubin 0.2-1.3 mg/dL
* Aspartate aminotransferase (AST) 0-35 U/L
* Alanine aminotransferase (ALT) 0-40 U/L
* Alkaline phosphatase 20-125 U/L
* Creatinine =< 1.2 mg/dL
* Potassium 3.5-5.0 mmol/L

Exclusion Criteria:

* Chronic medical illness, history of gastrointestinal disorders (e.g., ulcerative colitis, Crohn disease, celiac sprue, hereditary nonpolyposis colorectal cancer [HNPCC], familial adenomatous polyposis, pancreatic disease, previous gastrointestinal resection, radiation or chemotherapy, and cancer (other than non-melanoma skin cancer)
* Weight change greater than 4.5 kg within past year
* Oral or intravenous (IV) antibiotic use within the past 3 months
* Regular use of aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs)
* Smoking or use of cannabis products
* Known allergy to fish
* Intention to relocate out of study area within next 4 months

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Lampe, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fan YY, Salinas ML, Mullens DA, Davidson LA, Goldsby JS, Ivanov IV, Jayaraman A, Cai JJ, Levy L, Hullar MA, Navarro SL, Lampe JW, Chapkin RS. Pesco-Vegetarian Food Components Promote Colonocyte Froptosis in Preclinical Mouse Models and a Randomized Crossover Trial in Healthy Human Adults. J Nutr. 2025 Dec 27:101287. doi: 10.1016/j.tjnut.2025.101287. Online ahead of print. PMID 41461276

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred December 2020 thru March 2022 via ads, fliers and social media in the Seattle area. We received 243 screening questionnaires; 88 were incomplete. Of 155 completed, 95 were ineligible (61.3%). We contacted the 60 eligible; 43 attended orientation; 38 signed consent. Three were not randomized (2 ineligible based on abnormal clinical lab tests at baseline and 1 withdrew because of stool collection). Overall, we met planned recruitment goals.
Pre-assignment Details: Before randomization to determine the crossover order of supplements (active-washout-comparison, or comparison-washout-active), consented participants had a blood draw. Samples were sent to CLIA-certified Quest Labs for kidney/liver function tests as part of eligibility criteria. Two of the 38 were ineligible based on the lab test criteria. Additionally, 1 person decided they did not want to enter the trial and was not randomized.
Groups:
- Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator: Period 1: Fiber and Fish oil supplements (30 days) Washout: at least 60 days Period 2: Comparator supplements (30 days)
- Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil: Period 1: Comparator supplements (30 days) Washout: at least 60 days Period 2: Fiber and Fish oil supplements (30 days)
Period: Overall Study
Arm/Group | Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator | Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil
Started | 19 | 16
Completed Only Period 1 | 1 | 1
Completed (This total does not include the participants that only completed only study Period 1 and dropped out during the washout. The 2 participants who dropped out during the washout have partial measures (blood and stools) that may be included in some of the statistical analysis.) | 14 | 15
Not Completed | 5 | 1
Not completed — Withdrawal by Subject | 5 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator: Participants received a fiber supplement and fish oil supplement PO daily for 30 days. After a washout period, of at least 60 days, they received the comparator supplements (also for 30 days)
- Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil: Participants received the comparator supplements PO daily for 30 days. After a washout period, of at least 60 days, they received the fiber supplement and fish oil supplement (also for 30 days)
- Total: Total of all reporting groups
Arm/Group | Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator | Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (6.5) | 64.9 (5.3) | 62.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 15 | 15 | 30
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 12 | 14 | 26
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Feasibility and Retention for a Trial With Daily Doses of 35 g of Fiber and 6.2 g of EPA +DHA (and Corresponding Comparators)
Description: This grant is an R21 with the intent to provide preliminary data to propose a trial with a larger sample size and adequate statistical power.
Time Frame: Baseline to completion of the 2 study time periods
Population: All participants who consented and started the intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator: Period 1: participants receive fiber supplement and fish oil supplement PO daily on days 1-30.
  Washout: at least 60 days. Period 2: participants receive the comparators supplements also PO daily on days 90-120.
- Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil: For Period 1: participants receive comparator supplements PO daily on days 1-30.
  Participants enter a washout period for at least 60 days. For Period 2: participants receive fiber supplement and fish oil supplement also PO daily on days 90-120.
Arm/Group | Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator | Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil
Number analyzed (Participants) | 19 | 16
Participants
  Participants with complete measures (who completed Period 1 and Period 2) | 14 | 15
  Participants with partial measures (who only completed Period 1) | 1 | 1
  Participants who dropped out during Period 1 | 4 | 0
  Participants who dropped out during Period 2 | 0 | 0

2. Secondary Outcome: Number of Differentially Expressed Exfoliome Genes at p<0.01
Description: Poly A+ RNA was isolated from exfoliated cells in stool, and libraries generated from stool RNA and sequenced on an Illumina HiSeq 2500 platform. Intestinal exfoliome gene sequencing data from the end of each intervention period were analyzed using differential expression (DE) analysis. Count data were aligned, and sample libraries were filtered and normalized; 25,118 detected features were filtered to keep any feature with >20 cpm in 73% of samples in at least one of the groups; this resulted in 1000 genes. DE analysis between Fiber Plus Fish Oil Supplement vs the Comparator at the end time point was performed using edgeR with a paired design (Robinson et al, Bioinformatics 2010;26:139). Data are presented as number of DE genes significant at p < 0.01 (without multiple test correction). Upregulated genes indicate higher gene expression with Fiber Plus Fish Oil vs the Comparator and downregulated genes indicate lower gene expression with Fiber Plus Fish Oil vs the Comparator.
Time Frame: End of Fiber Plus Fish Oil Supplementation vs end of Comparator
Population: All participants who completed both the Fiber Plus Fish Oil Supplement and the Comparator intervention periods in this crossover study and had stools at the end of each intervention period were included in the analysis. RNA-Seq data from stool for 29 participants were analyzed for differential gene expression comparing the end of each intervention period.
Measure: Number; unit: number of genes at p<0.01
Units Other Than Participants: genes
Groups:
- Exfoliome Differentially Expressed (DE) Gene Analysis: Fiber plus fish oil supplementation vs comparator (based on end of treatment timepoints).
Arm/Group | Exfoliome Differentially Expressed (DE) Gene Analysis
Number analyzed (Participants) | 29
Number analyzed (genes) | 1000
number of genes at p<0.01
  Upregulated | 10
  Downregulated | 2
  Unchanged | 988

3. Secondary Outcome: Compliance
Description: Serum Phospholipids - Eicosapentaenoic acid (EPA), concentration
Time Frame: Average at the end of each intervention period
Measure: Mean (Standard Deviation); unit: mg/L
Groups:
- Fiber Plus Fish Oil Supplements: Daily Fiber plus Fish oil supplements (regardless of cross-over randomization order)
- Comparator: Daily comparator supplements
Arm/Group | Fiber Plus Fish Oil Supplements | Comparator
Number analyzed (Participants) | 31 | 31
mg/L | 43.9 (29.7) | 3.6 (3.0)

ADVERSE EVENTS:
Time Frame: Only during study participation (4 months)
Groups:
- Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator: Period 1: participants receive fiber supplement and fish oil supplements PO daily on days 1-30.
  Washout: at least 60 days. Period 2: participants receive the comparators supplements also PO daily on days 90-120.
- Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil: Period 1: participants receive the comparators supplements PO daily on days 1-30.
  Washout: at least 60 days. Period 2: participants receive fiber supplement and fish oil supplements also PO daily on days 90-120.
Arm/Group | Cross-over Randomization 1: Fiber Plus Fish Oil Followed by Comparator | Cross-over Randomization 2: Comparator Followed by Fiber Plus Fish Oil
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16

LIMITATIONS AND CAVEATS:
This is a pilot study with limited funding (R21 mechanism) thus sample size is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT04211766/Prot_SAP_001.pdf
  • Informed Consent Form (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/66/NCT04211766/ICF_000.pdf